CLINICAL TRIAL: NCT00408668
Title: Assessment of Protection Against Malaria by Sporozoite Challenge of Healthy Adults Vaccinated With the Virosomal Vaccine PEV3A and FP9-MVA ME-TRAP. A Phase I / IIa Controlled Challenge Trial
Brief Title: Efficacy of Combined PEV3A Virosomal Vaccine and FP9-MVA ME-TRAP Prime Boost Regimen
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council (Other Government); Pevion Biotech Ltd (Industry); Swiss Tropical & Public Health Institute (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC030; MRC agreement ID 74636
Record Dates: First submitted 2006-12-05; First posted 2006-12-07 (Estimated); Last update posted 2006-12-07 (Estimated); Status verified 2006-10

CONDITIONS: Malaria; Malaria, Falciparum
Keywords: Malaria Vaccine
MeSH Terms: conditions — Malaria; Malaria, Falciparum

INTERVENTIONS:
Biological: PEV3A
Biological: FP9 ME-TRAP
Biological: MVA ME-TRAP

SUMMARY:
The purpose of this study is to test three candidate malaria vaccines in new combinations to assess their efficacy at preventing malaria infection and triggering immune responses against malaria.

DETAILED DESCRIPTION:
Two of the vaccines ('FP9 ME-TRAP' and 'MVA ME-TRAP') have been designed at the University of Oxford. The other vaccine (PEV3A) has been designed jointly between the Swiss Tropical Institute and a Swiss company called Pevion Biotech Ltd. These are new vaccines that have been given to only a limited number of people before.

We aim to test these vaccines by:

* assessing their ability to prevent malaria infection
* determining how good they are at triggering a detectable immune response against malaria
* studying their safety further

Volunteers will be given up to six vaccinations over three months and will then be exposed to malaria infection. We do this by allowing mosquitoes infected with malaria to bite them under closely regulated conditions and observing if and when they develop blood stage malaria. If the vaccines provide some protection from malaria infection then either they will not develop malaria after the bites or the time taken to develop malaria will be longer. If not all volunteers are protected then we will be able to try and improve our vaccines by comparing the immune responses of volunteers who are protected to those not protected.

The information we get from this study may help to prevent malaria infection and disease in those who live in endemic areas and in travellers. The results of this study will be published in scientific journals and may be presented at professional meetings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Written informed consent
* Resident in or near Oxford for the duration of the vaccination study
* For women only, willingness to practice continuous effective contraception during the study and (if participating) during the subsequent challenge study.
* Agreement to refrain from blood donation during the course of the study
* Willingness to undergo an HIV test

Exclusion Criteria:

* Any deviation from the protocol defined normal range in biochemistry or haematology blood tests or in urine analysis
* Prior receipt of an investigational malaria vaccine
* Use of any investigational or non-registered drug, vaccine or medical device other than the study vaccine within 30 days preceding dosing of study vaccine, or planned use during the study period
* Administration of chronic immunosuppressive drugs or other immune modifying drugs within six months of vaccination.
* History of malaria chemoprophylaxis with chloroquine within 5 months prior to the planned challenge, with Lariam within 6 weeks prior to the challenge, and Riamet® within 2 weeks prior to the challenge
* Any history of malaria
* Travel to a malaria endemic area within the previous 6 months
* Planned travel to malarious areas during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection and asplenia
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of haemoglobinopathies
* History of diabetes mellitus
* Chronic or active neurological disease
* History of > 2 hospitalisations for invasive bacterial infections
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Hepatomegaly, right upper quadrant abdominal pain or tenderness
* Evidence of serious psychiatric condition
* Any on-going chronic illness requiring hospital specialist supervision
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Pregnant or lactating woman
* Any woman who is willing or intends to become pregnant during the study
* Any history of anaphylaxis in reaction to vaccination
* Principal Investigator assessment of lack of willingness to participate and comply with all requirements of the protocol
* History or clinical evidence of intravenous drug abuse
* Any other finding which in the opinion of the investigator would significantly increase the risk of having an adverse outcome from participating in this protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2005-08; Study Completion 2006-02

PRIMARY OUTCOMES:
Vaccine efficacy: The primary outcome is protection against malaria infection in a P. falciparum sporozoite challenge model.

SECONDARY OUTCOMES:
Immunogenicity - Vaccine immunogenicity assessed by IFN-γ ELISPOT and ELISA for vaccine specific antibodies
Safety - Vaccine safety assessed by collection of local and systemic adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, MA, BM BCh, DPhil, DM, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Thompson FM, Porter DW, Okitsu SL, Westerfeld N, Vogel D, Todryk S, Poulton I, Correa S, Hutchings C, Berthoud T, Dunachie S, Andrews L, Williams JL, Sinden R, Gilbert SC, Pluschke G, Zurbriggen R, Hill AV. Evidence of blood stage efficacy with a virosomal malaria vaccine in a phase IIa clinical trial. PLoS One. 2008 Jan 30;3(1):e1493. doi: 10.1371/journal.pone.0001493. PMID 18231580